CLINICAL TRIAL: NCT01469637
Title: A Phase 1, Randomized, Open-label, Crossover, Drug Interaction Study Evaluating the Pharmacokinetic Profiles of Sulfamethoxazole Administered Alone and in Combination With MMX® Mesalazine/Mesalamine in Healthy Adult Subjects
Brief Title: Sulfamethoxazole Drug Interaction Study With MMX® Mesalazine/Mesalamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPD476-117
Record Dates: First submitted 2011-11-04; First posted 2011-11-10 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — Sulfamethoxazole; Mesalamine

ARMS (2):
- Sulfamethoxazole + MMX placebo (Experimental)
  Interventions: Drug: sulfamethoxazole + MMX placebo
- Sulfamethoxazole + MMX Mesalazine/mesalamine (Experimental)
  Interventions: Drug: Sulfamethoxazole + MMX Mesalazine/mesalamine

INTERVENTIONS:
Drug: sulfamethoxazole + MMX placebo — 800 mg sulfamethoxazole/160 mg trimethoprim twice daily (BID) + MMX Mesalazine/mesalamine placebo once daily (QD) orally for 3 days, then a single dose of 800 mg sulfamethoxazole/160 mg trimethoprim + single does of MMX Mesalazine/mesalamine placebo orally on Day 4.
  Arms: Sulfamethoxazole + MMX placebo
Drug: Sulfamethoxazole + MMX Mesalazine/mesalamine — 800 mg sulfamethoxazole/160 mg trimethoprim BID + 4.8 g MMX Mesalazine/mesalamine QD for 3 days, then a single dose of 800 mg sulfamethoxazole/160 mg trimethoprim + a single dose of 4.8 g MMX Mesalazine/mesalamine on Day 4
  Other Names: Lialda
  Arms: Sulfamethoxazole + MMX Mesalazine/mesalamine

SUMMARY:
This is a drug interaction study evaluating the pharmacokinetic profiles of Sulfamethoxazole administered alone & in combination with Multi MatriX system (MMX®) formulation of mesalazine/mesalazine (Lialda®; Mesavancol®; Mezavant®) (MMX Mesalazine/mesalamine).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 years inclusive at the time of consent. The date of signing informed consent is defined as the beginning of the Screening Period.
2. Subject is willing to comply with any applicable contraceptive requirements of the protocol and is:

   * Male, or
   * Non-pregnant, non-lactating female
   * Females must be at least 90 days post-partum or nulliparous.

Exclusion Criteria

1. A history of current or recurrent disease that could affect the colon. This includes gastrointestinal disease, peptic ulceration, gastrointestinal bleeding, celiac disease, lactose intolerance, ulcerative colitis, Crohn's disease, or Irritable Bowel Syndrome. Subjects who have a history of chronic constipation, which is physician diagnosed and treated, will also be excluded from the study (frequency of bowel movements >48 hours between samples).
2. A history of current or relevant serious, severe, or unstable (acute or progressive) physical or psychiatric illness.
3. A history of gastrointestinal surgery performed within the past 12 months prior to the first dose of investigational product, with the exception of an appendectomy.
4. A history of or current clinically relevant moderate or severe renal or hepatic impairment.
5. A history of asthma or bronchospasm associated with the use of 5-ASA or other non-steroidal anti-inflammatory drugs.
6. Known or suspected intolerance or hypersensitivity to the investigational product or sulfamethoxazole/trimethoprim, closely related compounds, or any of the stated ingredients
7. A history of, or current, pancreatitis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-11-07 (Actual); Primary Completion 2011-12-20 (Actual); Study Completion 2011-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- PRA Inrernational, Lenexa, Kansas, United States

REFERENCES:
- [Derived] Pierce D, Corcoran M, Martin P, Barrett K, Inglis S, Preston P, Thompson TN, Willsie SK. Effect of MMX(R) mesalamine coadministration on the pharmacokinetics of amoxicillin, ciprofloxacin XR, metronidazole, and sulfamethoxazole: results from four randomized clinical trials. Drug Des Devel Ther. 2014 May 14;8:529-43. doi: 10.2147/DDDT.S55373. eCollection 2014. PMID 24868146

RESULTS

PARTICIPANT FLOW:
Groups:
- Sulfamethoxazole + MMX Placebo First: 800 mg sulfamethoxazole/160 mg trimethoprim twice daily (BID) + MMX placebo once daily (QD) orally for 3 days and a single dose of 800 mg sulfamethoxazole/160 mg trimethoprim + single does of MMX placebo orally on Day 4 for first intervention; then 800 mg sulfamethoxazole/160 mg trimethoprim BID + 4.8 g MMX Mesalazine/mesalamine QD for 3 days and a single dose of 800 mg sulfamethoxazole/160 mg trimethoprim + a single dose of 4.8 g MMX Mesalazine/mesalamine on Day 4 for second intervention.
- Sulfamethoxazole + MMX Mesalazine/Mesalamine First: 800 mg sulfamethoxazole/160 mg trimethoprim BID + 4.8 g MMX Mesalazine/mesalamine QD for 3 days and a single dose of 800 mg sulfamethoxazole/160 mg trimethoprim + a single dose of 4.8 g MMX Mesalazine/mesalamine on Day 4 for first intervention; then 800 mg sulfamethoxazole/160 mg trimethoprim twice daily (BID) + MMX placebo once daily (QD) orally for 3 days and a single dose of 800 mg sulfamethoxazole/160 mg trimethoprim + single does of MMX placebo orally on Day 4 for second intervention.
Period: First Intervention
Arm/Group | Sulfamethoxazole + MMX Placebo First | Sulfamethoxazole + MMX Mesalazine/Mesalamine First
Started | 22 | 22
Completed | 22 | 21
Not Completed | 0 | 1
Not completed — Unacceptable behavior | 0 | 1
Period: Second Intervention
Arm/Group | Sulfamethoxazole + MMX Placebo First | Sulfamethoxazole + MMX Mesalazine/Mesalamine First
Started | 22 | 21
Completed | 21 | 21
Not Completed | 1 | 0
Not completed — Incarcerated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulfamethoxazole + MMX Placebo First | Sulfamethoxazole + MMX Mesalazine/Mesalamine First | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (11.7) | 35.4 (12.6) | 36.7 (12.0)
Age, Customized [Count of Participants; unit: Participants]
  18 to 55 years of age | 22 | 22 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 12 | 12 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Within a Dosing Interval at Steady-State (AUCss) for Sulfamethoxazole
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure of how much and how long a drug stays in a body.
Time Frame: Assessed over a 24-hour period starting post-dose on day 4
Population: Pharmacokinetic Analysis Set defined as all subjects in the Safety Analysis Set for whom the primary pharmacokinetic data were considered sufficient and interpretable. Safety Analysis Set defined as subjects who took at least 1 dose of investigational product and had at least 1 postdose safety assessment.
Measure: Mean (Standard Deviation); unit: h*ug/ml
Groups:
- Sulfamethoxazole + MMX Placebo: 800 mg sulfamethoxazole/160 mg trimethoprim twice daily (BID) + MMX placebo once daily (QD) orally for 3 days and a single dose of 800 mg sulfamethoxazole/160 mg trimethoprim + single does of MMX placebo orally on Day 4.
- Sulfamethoxazole + MMX Mesalazine/Mesalamine: 800 mg sulfamethoxazole/160 mg trimethoprim BID + 4.8 g MMX Mesalazine/mesalamine QD for 3 days and a single dose of 800 mg sulfamethoxazole/160 mg trimethoprim + a single dose of 4.8 g MMX Mesalazine/mesalamine on Day 4.
Arm/Group | Sulfamethoxazole + MMX Placebo | Sulfamethoxazole + MMX Mesalazine/Mesalamine
Number analyzed (Participants) | 43 | 43
h*ug/ml | 786 (169) | 909 (198)
Statistical Analysis 1: Comparison: Sulfamethoxazole + MMX Placebo vs Sulfamethoxazole + MMX Mesalazine/Mesalamine; Test type: Non-Inferiority or Equivalence — If the 90% Confidence Intervals of the geometric mean ratio are wholly contained within the interval (0.80, 1.25), then the hypothesis of a drug interaction will be rejected; ANOVA; Geometric Mean ratio = 1.15, 90% CI 2-sided [1.12 to 1.18]

2. Primary Outcome: Maximum Plasma Concentration at Steady-State (Cmaxss) for Sulfamethoxazole
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: Assessed over a 24-hour period starting post-dose on day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Sulfamethoxazole + MMX Placebo | Sulfamethoxazole + MMX Mesalazine/Mesalamine
Number analyzed (Participants) | 43 | 43
ug/ml | 89.1 (16.3) | 100 (20.2)
Statistical Analysis 1: Comparison: Sulfamethoxazole + MMX Placebo vs Sulfamethoxazole + MMX Mesalazine/Mesalamine; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Mean Ratio = 1.12, 90% CI 2-sided [1.09 to 1.15]

ADVERSE EVENTS:
Arm/Group | Sulfamethoxazole + MMX Placebo | Sulfamethoxazole + MMX Mesalazine/Mesalamine
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 10/43 | 14/44
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulfamethoxazole + MMX Placebo (N=43) | Sulfamethoxazole + MMX Mesalazine/Mesalamine (N=44)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.